CLINICAL TRIAL: NCT04233463
Title: The Effect of Oral Polymeric Diet Enriched With TGF-beta 2 (Modulen) on Clinical Response and Mucosal Healing in Adult Patients With Newly Diagnosed Crohn's Disease: a Prospective, Randomized Study
Brief Title: The Effect of Oral Polymeric Diet Enriched With TGF-beta 2 (Modulen) on Clinical Response and Mucosal Healing in Adult Patients With Newly Diagnosed Crohn's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0128-18-HYMC
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modulen Diet (Active Comparator): Crohn patients will be given Modulen, an oral polymeric diet enriched with TGF-beta 2, along with a tailored diet
  Interventions: Dietary Supplement: Modulen
- Budesonide Treatment (Active Comparator): Crohn patients will be given Budesonide treatment
  Interventions: Drug: Budesonide

INTERVENTIONS:
Dietary Supplement: Modulen — Crohn patients will be given Modulen, an oral polymeric diet enriched with TGF-beta 2, along with a tailored diet
  Arms: Modulen Diet
Drug: Budesonide — Standard treatment for mild Crohn Disease patients
  Arms: Budesonide Treatment

SUMMARY:
The aim of this study is to evaluate prospectively a possible effect of an oral polymeric diet enriched with TGF-beta 2 (Modulen) as compared to Budesonide (one of the commonly accepted treatments for Crohn's disease) on clinical response, mucosal healing and intestinal microbiota in adult patients with newly diagnosed Crohn's disease using a capsule endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Crohn's Disease
* Mild to moderate severity

Exclusion Criteria:

* Patients who received systemic steroid or Budesonide or biological treatment
* Recent bowel surgery
* Colostomy, ileostomy
* Short bowel syndrome
* Obstructive symptoms
* Pregnancy, lactation
* Cardiac pacemaker or defibrillator
* Swallowing problems
* Uncontrolled metabolic diseases or any other condition that can be exacerbated by steroids

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Modulen Diet | 8 weeks
  Patients will undergo capsular endoscopy before and after dietary intervention and mucosal healing will be accessed using standard Lewis Score. Outcome will be compared to efficacy of Budesonide treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Baruch Ovadia, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No